CLINICAL TRIAL: NCT04318834
Title: Comprehensive Molecular Profiling of Advanced Biliary Tract Cancers for Better Treatment Selection: a McGill University Health Centre Study (COMPASS-B-MUHC)
Brief Title: Molecular Profiling of Advanced Biliary Tract Cancers
Acronym: COMPASS-B-MUHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Cancer Research Society (Other)
Responsible Party: Principal Investigator, George Zogopoulos, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-6112
Record Dates: First submitted 2020-02-24; First posted 2020-03-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary tract cancer; Cholangiocarcinoma; Molecular Profiling; Whole Genome Sequencing; Whole Transcriptome Sequencing
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with advanced biliary tract cancer (Experimental): Following a tumour biopsy for molecular profiling, chemo-naive patients with advanced biliary tract cancer will receive first-line gemcitabine-based chemotherapy or an investigational drug on a participating clinical trial.
  Interventions: Other: Tumour and germline molecular profiling

INTERVENTIONS:
Other: Tumour and germline molecular profiling — Tumour whole genome sequencing, germline whole genome sequencing, tumour whole transcriptome sequencing

SUMMARY:
Biliary tract cancer (BTC) accounts for <1% of all cancers, but remains a highly fatal malignancy. Surgical resection is the only hope for cure, but most patients present with advanced disease when curative-intent surgery is not possible. The therapeutic options for patients with advanced disease are limited, primarily to chemotherapeutic regimens, which are based on empiric evidence without the use of biomarkers. These current treatment strategies have been largely ineffective in controlling the disease, resulting in poor survival outcomes of less than 1 year. An understanding of the molecular characteristics of biliary tract cancer may enable stratification of patients into therapies that target specific molecular alterations with greater efficacies and improved clinical outcomes. This study aims to investigate the feasibility and clinical utility of prospective molecular profiling of advanced biliary tract cancer. The primary endpoint of this study is to demonstrate the feasibility of returning whole genome sequencing results within 8 weeks of tumour biopsy for second-line treatment consideration (n=30 patients). In parallel, tumour whole transcriptome sequencing will be performed to identify actionable molecular alterations (e.g., fusion transcripts). Once the primary endpoint is met, the study will be expanded. Current funding allows expansion to 40 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or radiological diagnosis of inoperable or metastatic BTC.
* Patient must have a tumour that is amenable to a core needle biopsy.
* Patients must have a measurable lesion by RECIST 1.1 in addition to the lesion that is going to be biopsied.
* Patients must be fit to safely undergo a tumour biopsy as judged by the investigator.
* Eastern Cooperative Group (ECOG) performance status ≤ 1.
* Life expectancy of greater than 90 days.
* Within 14 days of the proposed biopsy date, patients must have normal organ and marrow function.
* Patients must undergo systemic treatment with gemcitabine-based regimens as first-line standard systemic palliative treatment with or without other investigational agents within a clinical trial.
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients with one or more contraindications to tumour biopsy.
* Patients who have had any prior chemotherapy or other anti-cancer agent in the advanced stage setting.
* Patients who are currently on anti-cancer treatment.
* Patients with known brain metastases.
* Uncontrolled concurrent illness that would limit compliance with study requirements.
* Any other condition that would contraindicate the patient's participation due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tumour whole genome sequencing returned within 8 weeks | 2 years
  We have estimated that 30 patients will be required to reach the primary end point, which will be met if we demonstrate that tumor whole genome sequencing data is available at 8 weeks from the tumour biopsy for 80% of patients.

SECONDARY OUTCOMES:
Disease control rate | 4 years
  Number of patients that achieve stability of disease (cancer) by imaging (RECIST criteria) with first-line standard chemotherapy, consisting of gemcitabine backbone.
Progression-free survival rate | 4 years
  Progression free survival (PFS) defined as the interval between the date of registration and the earliest date of disease progression or death due to any cause of patients treated with 1st line chemotherapy.
Overall survival rate | 4 years
  Overall survival (OS) defined as the interval between the date of registration and the date of death of patients treated with 1st line chemotherapy.
Number of patients in whom at least 1 actionable mutation is identified | 4 years
  based on whole genome sequencing or RNA sequencing analyses.
Number of patients who received a targeted therapy (after first-line treatment) | 4 years
  based on the identification of an actionable mutation by whole genome sequencing or RNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No